CLINICAL TRIAL: NCT00004934
Title: A Randomized Trial of Paclitaxel/Epirubicin/Carboplatin Combination (TEC) Versus Paclitaxel/Carboplatin (TC) in the Treatment of Women With Advanced Ovarian Cancer
Brief Title: Paclitaxel and Carboplatin With or Without Epirubicin in Treating Patients With Stage IIB, Stage III, or Stage IV Invasive Ovarian Epithelial, Fallopian Tube, or Peritoneal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nordic Society of Gynaecological Oncology - Clinical Trials Unit (Other)
Collaborators: European Organisation for Research and Treatment of Cancer - EORTC (Network); NCIC Clinical Trials Group (Network)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000067620; NSGO-OC9804; CAN-NCIC-OV14; EORTC-55981
Record Dates: First submitted 2000-03-07; First posted 2003-01-27 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2003-05

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; fallopian tube cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Carboplatin; Epirubicin; Paclitaxel

INTERVENTIONS:
Drug: carboplatin
Drug: epirubicin hydrochloride
Drug: paclitaxel
Procedure: conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known whether receiving paclitaxel and carboplatin with epirubicin is more effective than paclitaxel and carboplatin alone for ovarian epithelial, fallopian tube, or peritoneal cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of paclitaxel and carboplatin with or without epirubicin in treating patients who have stage IIB, stage III, or stage IV invasive ovarian epithelial, fallopian tube, or peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare progression free survival and overall survival in patients with stage IIB, III, or IV invasive ovarian epithelial, fallopian tube, or peritoneal cancer treated with paclitaxel and carboplatin with or without epirubicin.
* Compare the toxicity of these 2 regimens in these patients.
* Compare the quality of life of patients treated with these 2 regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified by center and type of surgery (delayed surgery: 3 courses of chemotherapy before surgery vs primary surgery: optimally debulked stage IIB or III [residual tumor less than 1 cm] vs primary surgery: suboptimally debulked stage IV [residual tumor 1 cm or greater]).

Surgery

* Patients are assigned to one of two surgery groups:
* Group A: Patients undergo primary surgery comprised of hysterectomy, bilateral salpingo-oophorectomy (BSO), omentectomy, and resection of all tumor masses, if possible, before beginning chemotherapy. Patients with residual disease greater than 1 cm after completion of primary surgery receive 3 courses of chemotherapy, followed within 6 weeks by interval debulking surgery, followed within 3 weeks by the fourth course of chemotherapy.
* Group B: Patients undergo delayed surgery comprised of hysterectomy, BSO, omentectomy, and resection of all tumor masses, if possible, after completion of 3 courses of chemotherapy.

Chemotherapy

* Patients are randomized to 1 of 2 chemotherapy arms:
* Arm I: Patients receive epirubicin IV over 15-20 minutes, paclitaxel IV over 3 hours, and carboplatin IV over 1 hour on day 1. Treatment repeats every 3 weeks for 6 courses. Patients with residual tumor after completion of 6 courses may receive 3 additional courses.
* Arm II: Patients receive paclitaxel and carboplatin as above but no epirubicin. Quality of life is assessed before beginning study, after completion of courses 3, 6, and 9 (if applicable), and then at 6 and 12 months after completion of study treatment.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 800 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven stage IIB, III, or IV invasive ovarian epithelial, fallopian tube, or peritoneal cancer
* No symptomatic brain metastasis

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* WHO/ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,000/mm^3
* Neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 2 times upper limit of normal

Renal:

* Glomerular filtration rate at least 50 mL/min

Cardiovascular:

* No ventricular arrhythmia (LOWN class II or worse)
* No myocardial infarction within the past year
* No severe or uncontrolled hypertension
* No history of congestive heart disease (no New York Heart Association class III or IV heart disease) even if medically controlled
* LVEF at least 50%

Other:

* No other primary malignancies except carcinoma in situ of the cervix or basal cell skin cancer
* No worse than grade I preexisting motor or sensory neurologic pathology or symptoms
* No active infection or other serious underlying medical condition that would prevent compliance
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy
* No other concurrent antineoplastic agents

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy

Surgery:

* Not specified

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-08; Study Completion 2003-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar B. Kristensen, MD, PhD, Study Chair — Norwegian Radium Hospital; Ignace B. Vergote, MD, PhD, Study Chair — University Hospital, Gasthuisberg; Gavin C.E. Stuart, MD, Study Chair — Tom Baker Cancer Centre - Calgary
Locations (18):
- St. Mary's/Duluth Clinic Cancer Center, Duluth, Minnesota, United States
- U.Z. Gasthuisberg, Leuven, Belgium
- Canada (5):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Cancer Care Ontario-Hamilton Regional Cancer Centre, Hamilton, Ontario
  - CHUS-Hopital Fleurimont, Fleurimont, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
- Denmark (2):
  - Aalborg Hospital, Aalborg
  - Odense University Hospital, Odense
- Shaare Zedek Medical Center, Jerusalem, Israel
- Italy (3):
  - Spedali Civili, Brescia
  - Istituto Nazionale per lo Studio e la Cura dei Tumori, Milano (Milan)
  - Ospedale di Circolo e Fondazione Macchi, Varese
- Medisch Spectrum Twente, Enschede, Netherlands
- Norwegian Radium Hospital, Oslo, Norway
- Portugal (2):
  - Hospitais da Universidade de Coimbra (HUC), Coimbra
  - Instituto Portugues de Oncologia de Francisco Gentil - Centro de Lisboa, Lisbon
- Institut d'Oncologia Corachan, Barcelona, Spain

REFERENCES:
- [Result] Kristensen GB, Vergote I, Stuart G, Del Campo JM, Kaern J, Lopez AB, Eisenhauer E, Aavall-Lundquist E, Ridderheim M, Havsteen H, Mirza MR, Scheistroen M, Vrdoljak E. First-line treatment of ovarian cancer FIGO stages IIb-IV with paclitaxel/epirubicin/carboplatin versus paclitaxel/carboplatin. Int J Gynecol Cancer. 2003 Nov-Dec;13 Suppl 2:172-7. doi: 10.1111/j.1525-1438.2003.13363.x. PMID 14656276
- [Result] Kristensen G, Vergote I, Stuart G, et al.: First line treatment of ovarian cancer FIGO stages IIb-IV with paclitaxel/epirubicin/carboplatin (TEC) vs. paclitaxel/carboplatin (TC). Interim results of an NSGO-EORTC-NCIC CTG Gynecological Cancer Intergroup phase III trial. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-805, 2002.
- [Result] Lindemann K, Christensen RD, Vergote I, Stuart G, Izquierdo MA, Kaern J, Havsteen H, Eisenhauer E, Ridderheim M, Lopez AB, Hirte H, Aavall-Lundquvist E, Vrdoljak E, Green J, Kristensen GB. First-line treatment of advanced ovarian cancer with paclitaxel/carboplatin with or without epirubicin (TEC versus TC)--a gynecologic cancer intergroup study of the NSGO, EORTC GCG and NCIC CTG. Ann Oncol. 2012 Oct;23(10):2613-2619. doi: 10.1093/annonc/mds060. Epub 2012 Apr 26. PMID 22539562
- [Result] Kristensen GB, Vergote I, Stuart G, et al.: First-line treatment of ovarian/tubal/peritoneal cancer FIGO stage IIB-IV with paclitaxel/carboplatin with or without epirubicin (TEC vs TC). A gynecologic cancer intergroup study of the NSGO, EORTC GCG, and NCIC CTG. Results on progression-free survival. [Abstract] Int J Gynecol Cancer 15 (Suppl 3): 221, 2005.
- [Result] Kristensen GB, Vergote I, Eisenhauer E, et al.: First line treatment of ovarian/tubal/peritoneal cancer FIGO stage IIb-IV with paclitaxel/carboplatin with or without epirubicin (TEC vs TC). A Gynecologic Cancer Intergroup study of the NSGO, EORTC GCG, and NCIC CTG. Results on progression free survival. [Abstract] J Clin Oncol 22 (Suppl 14): A-5003, 449s, 2004.